CLINICAL TRIAL: NCT07311122
Title: Comparison of Endocrine Therapy Plus Ovarian Function Suppression and Chemotherapy Based on 21-gene RS in Young Age (≤ 50) Women (CUSTOM): Multi-center Registry Study
Brief Title: Endocrine Therapy Base on 21-gene RS
Acronym: CUSTOM
Status: Not yet recruiting | Type: Observational
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Soong June Bae, Associate Professor, Gangnam Severance Hospital
Other Study IDs: KBCSG 38
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Hormone receptor-positive; Oncotype DX; Chemotherapy; Ovarian function suppression
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Oncotype DX — All patients received Oncotype DX test.

SUMMARY:
Among patients aged ≤50 years with hormone receptor-positive, HER2-negative breast cancer and pathologic nodal stage pN0-1-limited to those with an Oncotype DX® Recurrence Score (RS) of 11-25 for pN0 and ≤25 for pN1-, we will investigate the followings:

i) Real-world patterns of adjuvant therapy (systemic chemotherapy and endocrine therapy) and radiotherapy according to N stage and Oncotype DX® RS.

ii) Clinicopathologic characteristics of each patient subgroup by adjuvant treatment modality and RS category.

iii) Survival outcomes and independent prognostic factors according to RS. iv) Survival analyses by adjuvant treatment modality, stratified by RS category, clinical risk, and N stage.

Through these analyses, we aim to establish clinical evidence on whether endocrine therapy combined with ovarian function suppression (OFS) can substitute for adjuvant chemotherapy in HR+/HER2- patients with pN0-1 disease within the above RS ranges, and-if so-to define the patient subsets for whom this substitution is appropriate.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed breast cancer.
2. Age ≤50 years at initial diagnosis.
3. Premenopausal at diagnosis, defined as any of the following:

   A. History of menstruation within 6 months prior to diagnosis. B. Serum FSH < 30 mIU/mL. C. If criteria A or B are unavailable, women aged ≤50 years are considered premenopausal.
4. Underwent curative-intent breast cancer surgery between January 2012 and December 2021.
5. Pathologic tumor stage pT1-pT3 after surgery.
6. Pathologic nodal stage pN0-pN1 after surgery.
7. Hormone receptor-positive disease by immunohistochemistry (IHC): estrogen receptor (ER) and/or progesterone receptor (PR) positive (≥1% positive cells or Allred score ≥3).
8. HER2-negative disease per ASCO/CAP guidelines: IHC 0 or 1+; if IHC 2+, in situ hybridization (FISH or SISH) negative.
9. Oncotype DX® performed, meeting one of the following Recurrence Score (RS) ranges:

A. pN0: RS 11-25. B. pN1: RS ≤25.

Exclusion Criteria:

1. Evidence of distant (systemic) metastasis at diagnosis.
2. Postmenopausal status at diagnosis, defined as any of the following:

   A. Prior bilateral oophorectomy before the breast cancer diagnosis (considered postmenopausal).

   B. Prior unilateral oophorectomy alone is not considered postmenopausal (classified as premenopausal).

   C. Bilateral oophorectomy performed after breast cancer surgery for therapeutic purposes is not an exclusion; such patients will be categorized as having received ovarian function suppression (OFS).

   D. Serum FSH ≥ 30 mIU/mL.
3. Hormone receptor-negative or HER2-positive disease.
4. Insufficient or unclear data regarding the type of adjuvant therapy received.
5. History of another malignancy treated before the breast cancer diagnosis, except for thyroid cancer and non-melanoma skin cancer.
6. Bilateral breast cancer.
7. Receipt of neoadjuvant systemic therapy prior to surgery.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study included the patients aged ≤ 50 years with hormone receptor-positive, HER2-negative breast cancer and pathologic nodal stage pN0-1 and those with an Oncotype DX® Recurrence Score (RS) of 11-25 for pN0 and ≤25 for pN1.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
invasive disease-free survival | 5 years after breast cancer diagnosis